CLINICAL TRIAL: NCT01720134
Title: The Impact of Legally Enforced Embryo Transfer Policy (Belgian Law 2003) on Cumulative Delivery Rate.
Status: Completed | Type: Observational
Sponsor: KU Leuven (Other)
Responsible Party: Principal Investigator, Sophie Debrock, Prof. Dr, KU Leuven
Other Study IDs: S53562
Record Dates: First submitted 2012-10-25; First posted 2012-11-02 (Estimated); Last update posted 2017-03-30 (Actual); Status verified 2017-03

CONDITIONS: Impact of Legislation on Cumulative Delivery Rate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- after legislation 1st july 2003: 2003-2006
- before legislation 1st july 2003: 1999-2003

SUMMARY:
Multiple pregnancy (MP) is associated with significant fetomaternal complications and a high cost. The multiple pregnancy rate per cycle (MPR) of treatment with Assisted Reproductive Technology (ART) is 25 % or higher even in countries where ART is reimbursed, much higher than the 1% after natural conception, related to the number of embryos transferred, and preventable by single embryo transfer (SET). In Belgium, the laboratory costs for 6 fresh ART cycles are reimbursed for female patients younger than 43 with a Belgian insurance number since July 2003, but only if a limited number of embryos is transferred depending on female age and cycle rank. Although this policy has resulted in a significant reduction in the MPR after ART in Belgium from 24 % to 13 %, available data are cycle based and it is unknown if the cumulative delivery rate per patient is affected by this legislation. The aim of this study was to test the hypothesis that Belgian ART legislation since 2003, coupling lab reimbursement to restriced embryo transfer policy, has resulted in a reduced CDR when compared to the situation before 2003.

ELIGIBILITY:
Inclusion Criteria:

* patients with their first IVF/ICSI cycle

Exclusion Criteria:

* cycles without oocytes or sperm, oocyte reception cycles, embryo reception cycles, cycles with preimplantation genetic diagnosis/screening

Ages: 18 Years to 43 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: patients undergoing IVF/ICSI cycles
Sampling Method: Non-Probability Sample
Enrollment: 1258 (Actual)
Dates: Start 2010-09; Primary Completion 2012-06 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
cumulative delivery rate | 1999-2006

CONTACTS AND LOCATIONS:
Locations (1):
- Leuven University Fertility Center, Leuven, Belgium